CLINICAL TRIAL: NCT06506422
Title: SGLT2 Inhibition as a Therapeutic Strategy to Reverse Arterial Stiffening in Aging
Brief Title: Empagliflozin Reversal of Arterial StiffnEss in Aging
Acronym: ERASE-Aging
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Camila Manrique, MD, Professor of Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2097602
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aging; Arterial Stiffness
MeSH Terms: interventions — empagliflozin; Exercise

STUDY DESIGN:
Intervention Model Description: double-blinded randomized placebo control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin (Experimental): 10mg Empagliflozin daily for 12 weeks
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): 10mg Placebo daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10mg Empagliflozin daily for 12 weeks
  Other Names: Active
  Arms: Empagliflozin
Drug: Placebo — 10mg Placebo daily for 12 weeks
  Other Names: Inactive
  Arms: Placebo

SUMMARY:
Randomized placebo-controlled clinical trial in a cohort of males (n=40) and females (n=40), 60-80 years of age, with the hypothesis that SGLT2 inhibition with empagliflozin (10mg/day for 12 weeks) reduces aging-related arterial stiffening.

DETAILED DESCRIPTION:
The investigators will employ a double-blinded randomized placebo control trial to determine the effects of 12 weeks of sodium glucose co-transporter 2 (SGLT2) inhibition with empagliflozin (10 mg daily), or matching placebo. Empagliflozin has been shown to decrease cardiovascular events and arterial stiffness in different populations. Placebo will be included for comparison purposes as empagliflozin is not a standard therapy for aging-associated arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent
* 60 to 80 years of age at randomization (women must be postmenopausal defined as more than 1 year without menses)
* Stable anti-hypertensive medication regimen (if in use) for at least 90 days
* Evidence of arterial stiffening (defined as carotid-femoral PWV >/= 8 m/s) at the time of screening visit.

Exclusion Criteria:

* Diabetes
* BMI>/= 45kg/m2
* Known history of cardiovascular disease: heart failure, ischemic heart disease, peripheral artery disease or stroke
* Estimated glomerular filtration rate GFR < 29 mL/min
* Active cancer (excluding basal cell carcinoma or stage 1 squamous cell carcinoma of the skin)
* Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
* Use of hormone replacement therapy
* Body weight change ≥10% within the last 6 months
* Uncontrolled hypertension during screening visit (>180/110 mmHg)
* Symptomatic hypotension and/or a SBP <100 mmHg
* History of ketoacidosis
* High fall risk per assessment of study physician and/or safety officer at the time of screening (results must be abnormal for both fall risk assessments and orthostatic blood pressure measurements)
* Anticipated need of prolonged fasting
* History of recurrent UTIs or mycotic genital infections
* Following a low-carbohydrate diet (<20 grams/day)
* Participation in regular exercise > 3 days/week per week at a moderate or vigorous intensity
* Known sensitivity to nitrate medications

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Carotid Femoral Pulse Wave Velocity (cfPWV) | Baseline (day 0), Week 4, Week 8, Final (week 12)
  cfPWV is the gold standard non-invasive index of arterial stiffness. Transit time between carotid and femoral pressure waves is calculated using the foot-to-foot method. cfPWV is calculated as distance traveled by the pulse wave (i.e., femoral location-sternal notch minus sternal notch-carotid location) divided by pulse transit time. All the measurements will be done by the same blinded technician. The goal is to assess changes from baseline when compared to weeks 4,8, and 12 time points.
  Report

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No